CLINICAL TRIAL: NCT00101205
Title: A Phase I Trial of the Combination of Oxaliplatin (NSC 266046, IND 57004), Ifosfamide, and Etoposide in Recurrent or Refractory Pediatric Solid Tumors and Lymphomas
Brief Title: Oxaliplatin, Ifosfamide and Etoposide in Treating Young Patients With Recurrent or Refractory Solid Tumors or Lymphoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00075; NCI-2009-00075 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000405828; OXALET (Other: St. Jude Children's Research Hospital); 6634 (Other: CTEP); P30CA021765 (NIH)
Record Dates: First submitted 2005-01-07; First posted 2005-01-10 (Estimated); Last update posted 2014-02-24 (Estimated); Status verified 2013-04

CONDITIONS: Angioimmunoblastic T-cell Lymphoma; B-cell Childhood Acute Lymphoblastic Leukemia; B-cell Chronic Lymphocytic Leukemia; Childhood Burkitt Lymphoma; Childhood Diffuse Large Cell Lymphoma; Childhood Grade III Lymphomatoid Granulomatosis; Childhood Immunoblastic Large Cell Lymphoma; Childhood Nasal Type Extranodal NK/T-cell Lymphoma; Hepatosplenic T-cell Lymphoma; Intraocular Lymphoma; Noncutaneous Extranodal Lymphoma; Peripheral T-cell Lymphoma; Recurrent Childhood Acute Lymphoblastic Leukemia; Recurrent Childhood Anaplastic Large Cell Lymphoma; Recurrent Childhood Grade III Lymphomatoid Granulomatosis; Recurrent Childhood Large Cell Lymphoma; Recurrent Childhood Lymphoblastic Lymphoma; Recurrent Childhood Small Noncleaved Cell Lymphoma; Recurrent Cutaneous T-cell Non-Hodgkin Lymphoma; Recurrent Mycosis Fungoides/Sezary Syndrome; Recurrent/Refractory Childhood Hodgkin Lymphoma; Refractory Chronic Lymphocytic Leukemia; Refractory Hairy Cell Leukemia; Small Intestine Lymphoma; T-cell Childhood Acute Lymphoblastic Leukemia; T-cell Large Granular Lymphocyte Leukemia; Unspecified Childhood Solid Tumor, Protocol Specific
MeSH Terms: conditions — Immunoblastic Lymphadenopathy; Leukemia, Lymphocytic, Chronic, B-Cell; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Extranodal NK-T-Cell; Intraocular Lymphoma; Lymphoma, T-Cell, Peripheral; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Large-Cell, Anaplastic; Dendritic Cell Sarcoma, Interdigitating; Lymphoma, T-Cell, Cutaneous; Mycosis Fungoides; Sezary Syndrome; Recurrence; Leukemia, Hairy Cell; Leukemia, Large Granular Lymphocytic | interventions — Oxaliplatin; Etoposide

ARMS (1):
- Arm I (Experimental): Patients receive oxaliplatin IV over 2 hours on day 1 and etoposide IV over 1 hour on days 1-3. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: oxaliplatin; Drug: etoposide

INTERVENTIONS:
Drug: oxaliplatin — Given IV
  Other Names: 1-OHP; Dacotin; Dacplat; Eloxatin; L-OHP
Drug: etoposide — Given IV
  Other Names: EPEG; VP-16; VP-16-213

SUMMARY:
This phase I trial is studying the side effects and best dose of oxaliplatin and etoposide in treating young patients with recurrent or refractory solid tumors or lymphomas. Drugs used in chemotherapy, such as oxaliplatin and etoposide, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Oxaliplatin may also help etoposide work better by making cancer cells more sensitive to the drug. Giving oxaliplatin together with etoposide may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the maximum tolerated dose of oxaliplatin and etoposide in pediatric patients with recurrent or refractory solid tumors or lymphoma.

II. Determine the dose-limiting toxic effects of this regimen in these patients.

SECONDARY OBJECTIVES:

I. Determine the pharmacokinetic profile of this regimen in these patients. II. Correlate the extent of oxaliplatin and etoposide exposure with toxic effects and therapeutic effects of this regimen in these patients.

III. Determine, preliminarily, the antitumor activity of this regimen in these patients.

OUTLINE: This is a dose-escalation study.

Patients receive oxaliplatin IV over 2 hours on day 1 and etoposide IV over 1 hour on days 1-3. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of oxaliplatin and etoposide until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Life expectancy > 8 weeks
* Albumin > 2 g/dL
* Histologically confirmed diagnosis of 1 of the following: solid tumor; histologic verification not required for brainstem tumors or optic pathway tumors; lymphoma; recurrent or refractory to conventional therapy OR no known effective therapy exists; bone marrow involvement allowed
* Performance Status: Karnofsky >= 50 % (patients > 10 years of age) OR Lansky >= 50% (patients for =< 10 years of age)
* Absolute neutrophil count > 1,000/mm^3
* Platelet count > 100,000/mm^3 (transfusion independent)
* Hemoglobin > 8 g/dL (transfusion allowed)
* ALT < 5.0 times ULN
* Creatinine normal OR glomerular filtration rate >= 80 mL/min/1.73 m^2
* Calcium normal (electrolyte supplements allowed)
* Echocardiogram and EKG normal
* Shortening fraction >= 27% OR ejection fraction > 50%
* No evidence of dyspnea at rest
* No exercise intolerance
* Pulse oximetry > 94% on room air
* Neurologic deficits due to CNS tumor must be relatively stable for >= 2 weeks before study entry
* Seizure disorder allowed provided well-controlled by non-enzyme-inducing anticonvulsants
* No peripheral neurotoxicity > grade 1
* Sodium, potassium, and magnesium normal (electrolyte supplements allowed)
* At least 1 week since prior biologic agents
* More than 1 week since prior growth factors
* More than 6 months since prior allogeneic peripheral blood stem cell transplantation AND no active graft-versus-host disease
* More than 3 weeks since prior myelosuppressive chemotherapy (6 weeks for nitrosoureas)
* More than 2 weeks since prior focal radiotherapy for symptomatic metastatic sites
* More than 6 weeks since prior substantial bone marrow radiotherapy
* More than 3 months since prior craniospinal (> 24 Gy), whole pelvis, or total-body radiotherapy
* Recovered from all prior therapy
* No concurrent enzyme-inducing anticonvulsants, including, but not limited to, the following: Barbiturates; Phenytoin; Carbamazepine

Exclusion Criteria:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No uncontrolled infection
* No history of life-threatening hypersensitivity to platinum-containing agents
* No prior oxaliplatin
* No other concurrent investigational agents
* No other concurrent anticancer therapy
* Inability or unwillingness of research participant or legal guardian/representative to give written informed consent.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2004-11; Primary Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
MTD of the combination of oxaliplatin and etoposide assessed by Common Terminology Criteria for Adverse Events (CTCAE) version 3.0 | 21 days
MTD of the addition of ifosfamide to the combination of oxaliplatin and etoposide assessed by CTCAE version 3.0 | 21 days

CONTACTS AND LOCATIONS:
Overall Officials: Lisa McGregor, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States